CLINICAL TRIAL: NCT00276939
Title: Plant-Based Dietary Intervention in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Diabetes Action Research and Education Foundation (Other); George Washington University (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCRM GWU DM Study
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Diet, Vegetarian; Diet, Fat-Restricted; Glycemic Index
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Fat-Restricted; Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Low-fat, low-Glycemic Index, vegan diet
  Interventions: Behavioral: Low-fat, low-Glycemic Index, vegan diet
- 2 (Active Comparator): ADA diet
  Interventions: Behavioral: Low-fat, low-Glycemic Index, vegan diet

INTERVENTIONS:
Behavioral: Low-fat, low-Glycemic Index, vegan diet

SUMMARY:
The purpose of the study is to assess whether, in individuals with type 2 diabetes, a low-fat, vegan diet improves blood glucose control more effectively than a control diet based on current American Diabetes Association (ADA) guidelines. The principal measure is hemoglobin A1c. Cardiovascular risk factors and dietary acceptability are also assessed. The study duration is 22 weeks with a one-year follow-up.

DETAILED DESCRIPTION:
Preliminary evidence suggests that low-fat, vegetarian regimens similar to those used to reverse coronary artery blockages may have a significant beneficial effect on type 2 diabetes, as demonstrated by reductions in fasting serum glucose concentrations and medication use. We therefore randomly assigned 99 individuals with type 2 diabetes to either a low-fat, vegan diet or a diet based on current American Diabetes Association guidelines for 22 weeks with a one-year follow-up period. The principal dependent measure is hemoglobin A1c. Cardiovascular risk factors are also being tracked, as is dietary acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus

Exclusion Criteria:

* hemoglobin A1c values <6.5% or >10.5%
* use of insulin for > 5 years
* tobacco use within the preceding 6 months
* consumption of more than 2 alcoholic beverages per day
* current drug abuse
* pregnancy
* unstable medical status
* current use of a low-fat, vegetarian diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 22 weeks

SECONDARY OUTCOMES:
Body weight | 22 weeks
Plasma lipid concentrations | 22 weeks
Urinary albumin | 22 weeks
Dietary Acceptability | 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Nicholson AS, Sklar M, Barnard ND, Gore S, Sullivan R, Browning S. Toward improved management of NIDDM: A randomized, controlled, pilot intervention using a lowfat, vegetarian diet. Prev Med. 1999 Aug;29(2):87-91. doi: 10.1006/pmed.1999.0529. PMID 10446033
- [Background] Barnard ND, Scialli AR, Turner-McGrievy G, Lanou AJ, Glass J. The effects of a low-fat, plant-based dietary intervention on body weight, metabolism, and insulin sensitivity. Am J Med. 2005 Sep;118(9):991-7. doi: 10.1016/j.amjmed.2005.03.039. PMID 16164885
- [Background] Jenkins DJ, Kendall CW, Marchie A, Jenkins AL, Augustin LS, Ludwig DS, Barnard ND, Anderson JW. Type 2 diabetes and the vegetarian diet. Am J Clin Nutr. 2003 Sep;78(3 Suppl):610S-616S. doi: 10.1093/ajcn/78.3.610S. PMID 12936955
- [Result] Barnard ND, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Jaster B, Seidl K, Green AA, Talpers S. A low-fat vegan diet improves glycemic control and cardiovascular risk factors in a randomized clinical trial in individuals with type 2 diabetes. Diabetes Care. 2006 Aug;29(8):1777-83. doi: 10.2337/dc06-0606. PMID 16873779
- [Result] Turner-McGrievy GM, Barnard ND, Cohen J, Jenkins DJ, Gloede L, Green AA. Changes in nutrient intake and dietary quality among participants with type 2 diabetes following a low-fat vegan diet or a conventional diabetes diet for 22 weeks. J Am Diet Assoc. 2008 Oct;108(10):1636-45. doi: 10.1016/j.jada.2008.07.015. PMID 18926128
- [Result] Barnard ND, Gloede L, Cohen J, Jenkins DJ, Turner-McGrievy G, Green AA, Ferdowsian H. A low-fat vegan diet elicits greater macronutrient changes, but is comparable in adherence and acceptability, compared with a more conventional diabetes diet among individuals with type 2 diabetes. J Am Diet Assoc. 2009 Feb;109(2):263-72. doi: 10.1016/j.jada.2008.10.049. PMID 19167953
- [Result] Barnard ND, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Green A, Ferdowsian H. A low-fat vegan diet and a conventional diabetes diet in the treatment of type 2 diabetes: a randomized, controlled, 74-wk clinical trial. Am J Clin Nutr. 2009 May;89(5):1588S-1596S. doi: 10.3945/ajcn.2009.26736H. Epub 2009 Apr 1. PMID 19339401
- [Result] Barnard ND, Noble EP, Ritchie T, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Green AA, Ferdowsian H. D2 dopamine receptor Taq1A polymorphism, body weight, and dietary intake in type 2 diabetes. Nutrition. 2009 Jan;25(1):58-65. doi: 10.1016/j.nut.2008.07.012. Epub 2008 Oct 2. PMID 18834717
- [Derived] Turner-McGrievy GM, Jenkins DJ, Barnard ND, Cohen J, Gloede L, Green AA. Decreases in dietary glycemic index are related to weight loss among individuals following therapeutic diets for type 2 diabetes. J Nutr. 2011 Aug;141(8):1469-74. doi: 10.3945/jn.111.140921. Epub 2011 Jun 8. PMID 21653575